CLINICAL TRIAL: NCT04464772
Title: FreeStyle Libre Continuous Glucose Monitoring System Accuracy Study
Status: Completed | Type: Observational
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC-US-VAL-20192
Record Dates: First submitted 2020-07-07; First posted 2020-07-09 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: FreeStyle Libre 3 — FreeStyle Libre 3 Continuous Glucose Monitoring System

SUMMARY:
The purpose of this study is to characterize the Freestyle Libre Glucose Monitoring System in pediatric and adult subjects with respect to YSI reference venous plasma sample measurements.

DETAILED DESCRIPTION:
Up to 100 subjects will be enrolled at up to six (6) clinical research sites in the United States. Subjects will wear two Sensors. Each Sensor will have a paired Reader that will be given to the subject. Subjects will be asked to perform at least 4 capillary Blood Glucose (BG) tests per day using the primary Reader.

Interstitial glucose readings from each Sensor will be obtained with the corresponding Readers immediately following each BG test. Subjects will be instructed to report any problems with the device. Subjects will make up to six (6) scheduled visits to the clinical study site, including the Enrollment/Screening Visit (Visit 1). Based on the subjects' age and

/or weight, subjects will have up to three (3) in- clinic visits during which intravenous blood draws and YSI reference testing will occur.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 4 years of age.
2. Subject must have type 1 or type 2 diabetes.
3. Subject must require insulin therapy through an insulin pump and/or multiple daily insulin injections (at least 3 injections daily).
4. Willing to perform a minimum of 4 finger sticks per day while wearing the sensor in the study.
5. Subject must be able to read and understand English.
6. For subjects age 6 and older: willing to allow medical personnel to insert an IV catheter in the arm to allow for venous blood samples to be obtained per the study protocol.
7. In the investigator's opinion, the subject must be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol.
8. At the time of enrollment, subject must be available to participate in all study visits.
9. Subjects aged 18 years and older must be willing and able to provide written signed and dated informed consent.
10. Subjects aged 17 years and younger must have a parent, guardian or legally authorized representative willing and able to provide written informed consent.
11. Subjects aged 7 - 17 years of age must be willing and able to provide written signed and dated informed assent.

Exclusion Criteria:

1. Subject has known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin.
2. Subjects age 18 and older: Subject is known to be pregnant, attempting to conceive or is not willing and able to practice birth control during the study duration (applicable to only to female subjects age 18 and older).
3. Subjects age 17 and younger: Subject is known to be pregnant or becomes pregnant during the study (only applicable to female subjects age 17 years and younger)
4. Subject has extensive skin changes/diseases at the proposed application sites that could interfere with device placement or the accuracy of interstitial glucose measurements. Such conditions include, but are not limited to extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, dermatitis herpetiformis, skin lesions, redness, infection or edema.
5. Subject is currently participating in another clinical trial.
6. Subject has donated blood within 112 days (3.7 months) prior to the beginning of the study activities.
7. For subjects age 6 and older: subject has a hemoglobin (Hb) level that is below the normal range (for reference the low end of the normal range for Hb for adult males is 14 g/dL and for adult females is 12 g/dL; for pediatric males and pediatric 13.0 g/dL; for pediatric females aged 12 - 17 it is 12.0 g/dL2).
8. Subject has a known concomitant medical condition which, in the opinion of the investigator, could present a risk to the safety or welfare of the subject or study staff.
9. Subject has X-ray, MRI, CT or diathermy appointment scheduled during the period of study participation, and the appointment cannot be rescheduled for a time before study participation starts or after study participation ends.
10. Subject is unsuitable for participation due to any other cause as determined by the Investigator.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric subjects with type 1 or type 2 diabetes requiring multiple daily insulin injections (MDI) or continuous subcutaneous insulin infusion (CSII).
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
System Performance | 45 days
  System Performance will be characterized with respect to YSI reference venous plasma measurements

CONTACTS AND LOCATIONS:
Overall Officials: Shridhara A Karinka, PhD, Study Director — Abbott Diabetes Care
Locations (4):
- United States (4):
  - AMCR Institute, Escondido, California
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Rocky Mountain Diabetes & Osteoporosis Center, Idaho Falls, Idaho
  - Rainier Clinical Research, Renton, Washington

IPD SHARING:
Plan to Share IPD: Undecided